CLINICAL TRIAL: NCT05333796
Title: The Effect of Back Muscles Activation on Idiopathic Scoliosis Using Surface Electromyography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-2203-747-302
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Scoliosis
MeSH Terms: interventions — Gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy children (5 to 12 years old) (Experimental)
  Interventions: Behavioral: gait with leg length discrepancy

INTERVENTIONS:
Behavioral: gait with leg length discrepancy — After attaching the surface electromyography(EMG) to bilateral back muscles, participants walk at a comfortable speed. The investigators will evaluate the effects of leg length discrepancy on the back muscle activation during gait.

SUMMARY:
The purpose of this study is to evaluate the effect of back muscle activations on idiopathic scoliosis

DETAILED DESCRIPTION:
* Design: Prospective study
* Setting: hospital rehabilitation department
* Intervention: Participants were asked to walk with a surface electromyography(EMG) attached to their back muscles. After repeating the same process with different leg lengths discrepancy (0cm, 0.5cm, 1cm), participants are compared the main outcome measures.
* Main outcome measures: surface electromyography(EMG)

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (5 to 12 years old)

Exclusion Criteria:

* Children with leg length discrepancy over 0.5cm
* Children complaining of acute low back pain
* Children with spinal scoliosis
* Children with cerebral palsy, muscle paralysis, polio, congenital spinal abnormalities
* Children who underwent spinal surgery

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
surface electromyography | 20 minutes
  surface muscle contraction of bilateral back muscles
  * bilateral spinal muscles on T6, T12, L3
  * bilateral quadratus lumborum muscles
  * bilateral iliopsoas muscles

CONTACTS AND LOCATIONS:
Overall Officials: Jusuk Ryu, M.D. PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea